CLINICAL TRIAL: NCT01096849
Title: A Double-blind, Randomized, Comparator-controlled Study to Assess the Safety, Efficacy, and Pharmacokinetics of ACHN-490 Injection Administered IV in Patients With Complicated Urinary Tract Infections or Acute Pyelonephritis
Brief Title: A Study of Plazomicin Compared With Levofloxacin for the Treatment of Complicated Urinary Tract Infection (cUTI) and Acute Pyelonephritis (AP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-490-002
Record Dates: First submitted 2010-03-12; First posted 2010-03-31 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
Keywords: urinary tract infection; UTI; cUTI; pyelonephritis; AP; ACHN-490
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — Levofloxacin; plazomicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- plazomicin (10 mg/kg) (Experimental): Patients received two intravenous (IV) infusions daily for 5 consecutive days: 10 milligrams per kilogram (mg/kg) plazomicin followed by placebo.
  Interventions: Drug: plazomicin; Drug: placebo
- plazomicin (15 mg/kg) (Experimental): Patients received two IV infusions daily for 5 consecutive days: 15 mg/kg plazomicin followed by placebo.
  Interventions: Drug: plazomicin; Drug: placebo
- levofloxacin (Active Comparator): Patients received two IV infusions daily for 5 consecutive days: placebo followed by 750 milligrams (mg) levofloxacin.
  Interventions: Drug: levofloxacin; Drug: placebo

INTERVENTIONS:
Drug: levofloxacin
  Arms: levofloxacin
Drug: plazomicin
  Arms: plazomicin (10 mg/kg); plazomicin (15 mg/kg)
Drug: placebo

SUMMARY:
This was a multi-center, multi-national, double-blind, randomized, comparator-controlled study of plazomicin administered intravenously compared with levofloxacin, a standard approved intravenous therapy for complicated urinary tract infection (cUTI) and acute pyelonephritis (AP).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented or suspected cUTI/AP with clinical signs and symptoms
* Normal kidney function defined as creatinine clearance (CLcr) of ≥60mL/min using Cockcroft-Gault formula

Key Exclusion Criteria:

* Acute bacterial prostatis, orchitis, epididymitis, or chronic bacterial prostatis
* Gross heanaturia requiring intervention other than study drug
* Urinary tract surgery within 7 days of randomization or during the study period
* A known nonrenal source of infection diagnosed within 7 days of randomization
* A corrected QT interval > 440 msec
* History of hearing loss with onset before the age of 40 years, sensorineural hearing loss, or family history of hearing loss
* Pregnant or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2012-04-03 (Actual); Study Completion 2012-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Achaogen, Inc.

REFERENCES:
- [Background] Connolly LE, Riddle V, Cebrik D, Armstrong ES, Miller LG. A Multicenter, Randomized, Double-Blind, Phase 2 Study of the Efficacy and Safety of Plazomicin Compared with Levofloxacin in the Treatment of Complicated Urinary Tract Infection and Acute Pyelonephritis. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e01989-17. doi: 10.1128/AAC.01989-17. Print 2018 Apr. PMID 29378708

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Started | 22 | 76 | 47
Completed | 20 | 64 | 41
Not Completed | 2 | 12 | 6
Not completed — Consent Withdrawn | 1 | 4 | 2
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Unacceptable/ Intolerable AE(s) | 0 | 1 | 1
Not completed — Investigator or Medical Monitor Decision | 0 | 1 | 0
Not completed — Administrative Reasons | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all randomized patients.
Groups:
- Plazomicin (10 mg/kg): Patients received two IV infusions daily for 5 consecutive days: 10 mg/kg plazomicin followed by placebo.
- Levofloxacin: Patients received two IV infusions daily for 5 consecutive days: placebo followed by 750 mg levofloxacin.
- Total: Total of all reporting groups
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin | Total
Number analyzed (Participants) | 22 | 76 | 47 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 72 | 42 | 131
  >=65 years | 5 | 4 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (18.12) | 40.00 (15.02) | 44.8 (14.61) | 42.6 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 61 | 37 | 116
  Male | 4 | 15 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Attained Microbiological Eradication (MBE) at the Test of Cure (TOC) Visit in the Microbiological Intent to Treat (MITT) Population
Description: MBE was defined as documented eradication of all isolated pathogens. This was based on a urine culture, taken at the TOC visit that showed that all pathogens isolated at baseline at ≥10^5 colony forming unit(s) per milliliter (CFU/mL) were reduced to <10^4 CFU/mL.
Time Frame: Day 1 to TOC (Day 12)
Population: The MITT population was defined as a subset patients from the ITT population with at least one isolated causative pathogen from an acceptable pretreatment urine specimen.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 12 | 51 | 29
percentage of patients | 50 [21.1 to 78.9] | 60.8 [46.1 to 74.2] | 58.6 [38.9 to 76.5]

2. Primary Outcome: Percentage of Patients Who Attained MBE at the TOC Visit in the Microbiologically Evaluable (ME) Population
Description: MBE was defined as documented eradication of all isolated pathogens. This was based on a urine culture, taken at the TOC visit that showed that all pathogens isolated at baseline at ≥10^5 CFU/mL were reduced to <10^4 CFU/mL.
Time Frame: Day 1 to TOC (Day 12)
Population: The ME population was defined as clinically evaluable (CE) patients who had a causative pathogen isolated at baseline (ie, patients in both the MITT and CE populations). To be included in the ME population, a patient must also have had results obtained from non-contaminated urine culture at TOC.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients | 85.7 [42.1 to 99.6] | 88.6 [73.3 to 96.8] | 81.0 [58.1 to 94.6]

3. Primary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered to be drug related. An AE (also referred to as an adverse experience) can be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, and it does not imply any judgment about causality. Adverse events also include the exacerbation or worsening of a condition present at screening other than the index infection for which the patient was enrolled in the study. A TEAE is any AE that newly appeared, increased in frequency, or worsened in severity following initiation of study drug.
Time Frame: Day 1 to the end of study (Day 40)
Population: The Safety population was defined as all randomized patients who received any amount of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 22 | 74 | 44
percentage of patients | 31.8 | 35.1 | 47.7

4. Secondary Outcome: Percentage of Patients Who Attained Clinical Cure Based on Investigator and Sponsor Assessments at TOC Visit in the Intent-to-treat (ITT) Population
Description: Investigator's assessment criteria defined Clinical Cure as resolution of baseline clinical signs and symptoms of infection through the TOC visit.
  The sponsor's assessment criteria was programmatically based on the investigator's assessment of participant clinical outcome, the number of days and doses of drug received and whether an antibiotic was administered.
Time Frame: Day 1 to TOC (Day 12)
Population: The intent-to-treat (ITT) population was defined as all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 22 | 76 | 47
percentage of patients
  Investigator's Assessment: Cured | 63.6 [40.7 to 82.8] | 69.7 [58.1 to 79.8] | 70.2 [55.1 to 82.7]
  Sponsor's Assessment: Cured | 59.1 [36.4 to 79.3] | 69.7 [58.1 to 79.8] | 68.1 [52.9 to 80.9]

5. Secondary Outcome: Percentage of Patients Who Attained Clinical Cure Based on Investigator and Sponsor Assessments at the TOC Visit in the CE Population
Description: Investigator's assessment criteria defined Clinical Cure as a resolution of baseline clinical signs and symptoms of infection through the TOC visit.
  The sponsor's assessment criteria was programmatically based on the investigator's assessment of participant clinical outcome, the number of days and doses of drug received and whether an antibiotic was administered.
Time Frame: Day 1 to TOC (Day 12)
Population: The CE population was defined as patients who received at least 80% of study drug for clinical successes or 40% for clinical failures and must not have had indeterminate clinical response at TOC.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 18 | 64 | 42
percentage of patients
  Investigator's Assessment: Cured | 66.7 [41.0 to 86.7] | 76.6 [64.3 to 86.2] | 78.6 [63.2 to 89.7]
  Sponsor's Assessment: Cured | 66.7 [41.0 to 86.7] | 76.6 [64.3 to 86.2] | 76.2 [60.5 to 87.9]

6. Secondary Outcome: Percentage of Patients Who Attained Clinical Cure Based on Investigator and Sponsor Assessments at the End of Treatment (EOT) Visit in the CE Population
Description: Investigator's assessment criteria defined Clinical Cure as a resolution of baseline clinical signs and symptoms of infection through the EOT visit.
  The Sponsor's assessment criteria was programmatically based on the investigator's assessment of participant clinical outcome, the number of days and doses of drug received and whether an antibiotic was administered.
Time Frame: Day 1 to EOT (Day 5)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 18 | 64 | 42
percentage of patients
  Investigator's Assessment: Cured | 94.4 [72.7 to 99.9] | 82.8 [71.3 to 91.1] | 88.1 [74.4 to 96.0]
  Sponsor's Assessment: Cured | 94.4 [72.7 to 99.9] | 82.8 [71.3 to 91.1] | 85.7 [71.5 to 94.6]

7. Secondary Outcome: Percentage of Patients Who Attained MBE at the EOT Visit in the ME Population
Description: MBE was defined as documented eradication of all isolated pathogens. This was based on a urine culture, taken at the EOT visit that showed that all pathogens isolated at baseline at ≥10^5 CFU/mL were reduced to <10^4 CFU/mL.
Time Frame: Day 1 to EOT (Day 5)
Population: The ME population was defined as CE patients who had a causative pathogen isolated at baseline (ie, patients in both the MITT and CE populations). To be included in the ME population, a patient must also have had results obtained from non-contaminated urine culture at TOC.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients | 85.7 [42.1 to 99.6] | 82.9 [66.4 to 93.4] | 76.2 [52.8 to 91.8]

8. Secondary Outcome: Percentage of Patients Who Attained MBE at the EOT Visit in the MITT Population
Description: as for outcome 7
Time Frame: Day 1 to EOT (Day 5)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 12 | 51 | 29
percentage of patients | 83.3 [51.6 to 97.9] | 74.5 [60.4 to 85.7] | 72.4 [52.8 to 87.3]

9. Secondary Outcome: Percentage of Patients Who Attained MBE at the TOC Visit in the ME Population by Baseline Pathogen
Description: as for outcome 2
Time Frame: Day 1 to TOC (Day 12)
Population: as for outcome 7
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients
  Gram-positive bacteria (aerobes), eradication | 100 | 100 | 100
  Gram-negative bacteria (aerobes), eradication | 83.3 | 87.5 | 80.0

10. Secondary Outcome: Percentage of Patients Who Attained MBE at the TOC Visit in the ME Population Stratified by Infection Category
Description: as for outcome 2
Time Frame: Day 1 to TOC (Day 12)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients
  Acute pyelonephritis, eradication: number analyzed (Participants) | 2 | 18 | 15
  Acute pyelonephritis, eradication | 100 [15.8 to 100.0] | 88.9 [65.3 to 98.6] | 80 [51.9 to 95.7]
  Complicated Lower UTI, eradication: number analyzed (Participants) | 5 | 17 | 6
  Complicated Lower UTI, eradication | 80.0 [28.4 to 99.5] | 88.2 [63.6 to 98.5] | 83.3 [35.9 to 99.6]
  cUTI with indwelling catheter, eradication: number analyzed (Participants) | 1 | 4 | 0
  cUTI with indwelling catheter, eradication | 0 [0 to 97.5] | 75 [19.4 to 99.4] |
  cUTI without indwelling catheter, eradication: number analyzed (Participants) | 4 | 13 | 6
  cUTI without indwelling catheter, eradication | 100 [39.8 to 100.0] | 92.3 [64.0 to 99.8] | 83.3 [35.9 to 99.6]

11. Secondary Outcome: Percentage of Patients Who Attained MBE at the TOC Visit in the ME Population by Country/Region
Description: as for outcome 2
Time Frame: Day 1 to TOC (Day 12)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients
  India, eradicaton: number analyzed (Participants) | 3 | 6 | 3
  India, eradicaton | 66.7 [9.4 to 99.2] | 66.7 [22.3 to 95.7] | 0 [0 to 70.8]
  Latin America, eradication: number analyzed (Participants) | 2 | 11 | 8
  Latin America, eradication | 100 [15.8 to 100] | 100 [71.5 to 100] | 100 [63.1 to 100]
  North America, eradication: number analyzed (Participants) | 2 | 18 | 10
  North America, eradication | 100 [15.8 to 100] | 88.9 [65.3 to 98.6] | 90 [55.5 to 99.7]

12. Secondary Outcome: Time (Days) to Resolution of Signs and Symptoms of cUTI and AP in the MITT Population
Description: Resolution of clinical signs and symptoms is defined as absence of all signs and symptoms present at baseline.
Time Frame: Day 1 to End of Study (Day 40)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 12 | 51 | 29
days | 11.8 (2.67) | 10.7 (1.93) | 13.3 (3.16)

13. Secondary Outcome: Time (Days) to Clinical Cure Based on Investigator's and Sponsor's Assessments in the MITT Population
Description: as for outcome 5
Time Frame: Day 1 to End of Study (Day 40)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 12 | 51 | 29
days
  Investigator's Assessment: number analyzed (Participants) | 8 | 39 | 20
  Investigator's Assessment | 9.5 (2.43) | 7.0 (0.71) | 7.6 (0.82)
  Sponsor's Assessment: number analyzed (Participants) | 8 | 39 | 19
  Sponsor's Assessment | 9.5 (2.43) | 7.0 (0.71) | 7.4 (0.83)

14. Secondary Outcome: Time (Days) to Defervescense in the MITT Population
Description: Defervescence is defined as the absence of fever <37.7 degrees Celsius and is assessed in patients who were afebrile at baseline.
Time Frame: Day 1 to End of Study (Day 40)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 1 | 9 | 3
days | 1.0 | 2.1 (0.26) | 2.0 (0.58)

15. Secondary Outcome: Percentage of Patients Experiencing a Clinical Relapse or Microbiological Recurrence in the ME Population
Description: Patients who had a clinical relapse (defined as the return of clinical signs and symptoms requiring antibiotic therapy) or microbiological recurrence (defined as eradication of the original pathogen[s] at the TOC visit but regrowth at the level >10^5 CFU/mL by the LTFU [long term follow up] visit).
Time Frame: Day 1 to LTFU (Day 40)
Population: as for outcome 7
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients
  Clinical Relapse | 0 | 14.3 | 6.3
  Microbiological Recurrence | 0 | 6.5 | 23.5

16. Secondary Outcome: Percentage of Patients With a Superinfection or New Infection in the ME Population
Description: Superinfections are defined as a pathogen other than the one at baseline found in urine at ≥10^5 CFU/mL any time after the first infusion through EOT. New infections are defined as a pathogen other than the one at baseline found in urine at ≥10^5 CFU/mL any time after EOT.
Time Frame: Day 1 to to End of Study (Day 40)
Population: as for outcome 7
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
Number analyzed (Participants) | 7 | 35 | 21
percentage of patients
  Superinfection | 28.6 | 8.6 | 0
  New infection | 0 | 2.9 | 4.8

ADVERSE EVENTS:
Time Frame: Day 1 to the end of the study (Day 40)
Description: The safety population, all randomized patients who received any amount of study drug.
Arm/Group | Plazomicin (10 mg/kg) | Plazomicin (15 mg/kg) | Levofloxacin
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/74 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/74 | 2/44
Other Adverse Events (participants affected / at risk) | 2/22 | 22/74 | 3/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plazomicin (10 mg/kg) (N=22) | Plazomicin (15 mg/kg) (N=74) | Levofloxacin (N=44)
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plazomicin (10 mg/kg) (N=22) | Plazomicin (15 mg/kg) (N=74) | Levofloxacin (N=44)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2
Nausea (Gastrointestinal disorders) | 0 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
Headache (Nervous system disorders) | 2 | 6 | 3
Dizziness (Nervous system disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may publish/present the study results provided all of the following: (i) the primary publication has been published; or, if no such publication has occurred, at least 18m have passed since the completion of the study; (ii) Achaogen is allowed at least 60d to review; (iii) confidential information is deleted as requested; (iv) comments and proposed revisions are considered; and (v) during the 60d review, if requested, the Investigator shall delay the publication or presentation.